CLINICAL TRIAL: NCT05108051
Title: A Phase 1, Open-Label, Three-Period, Single-center Study to Assess the Pharmacokinetic Interactions Between ZSP1273 and Oseltamivir in Healthy Subjects
Brief Title: Study to Investigate the Potential Drug-Drug Interaction Between ZSP1273 and Oseltamivir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ZSP1273-20-05
Record Dates: First submitted 2021-09-29; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — ZSP1273; Oseltamivir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sequence 1 (Experimental): Period 1: study of ZSP1273's pharmacokinetics at steady state； Period 2: study of Oseltamivir's pharmacokineticsat at steady state； Period 3: study of ZSP1273's pharmacokinetics under Oseltamivir at steady state.
  Interventions: Drug: ZSP1273; Drug: Oseltamivir
- sequence 2 (Experimental): Period 1: study of Oseltamivir's pharmacokineticsat at steady state; Period 2: study of ZSP1273's pharmacokinetics under Oseltamivir at steady state; Period 3: study of ZSP1273's pharmacokinetics at steady state.
  Interventions: Drug: ZSP1273; Drug: Oseltamivir
- sequence 3 (Experimental): Period 1: study of ZSP1273's pharmacokinetics under Oseltamivir at steady state; Period 2: study of ZSP1273's pharmacokinetics at steady state; Period 3: study of Oseltamivir's pharmacokineticsat at steady state.
  Interventions: Drug: ZSP1273; Drug: Oseltamivir

INTERVENTIONS:
Drug: ZSP1273 — ZSP1273 tablets 600mg administered orally once daily
Drug: Oseltamivir — Oseltamivir 75mg administered orally twice daily

SUMMARY:
To evaluate the drug-drug interaction between ZSP1273 and oseltamivir, the pharmacokinetic characteristics and safety of ZSP1273 and oseltamivir in healthy subjects, so as to provide a basis for the design of administration regimen in subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects between 18-45 years (Both inclusive);
* Body weight is no less than 50kg in males and no less than 45kg in females.Body mass index (BMI) 18~26 kg/m2 (Both inclusive); BMI is determined by the following equation: BMI = weight/height2 (kg/m2);
* Subjects (including partners) are willing to voluntarily use effective contraception from screening to 3 months after the last study drug administration.

Exclusion Criteria:

* Known history of allergic constitution (multiple drugs especially with ZSP1273 or oseltamivir and its preparation of the main ingredient allergy, food allergy);
* Subjects who donated blood or bleeding profusely(> 450 mL)in the 3 months preceding study screening;
* History or presence of any disease or condition known to increase the risk of bleeding, eg.hemorrhoids, acute gastritis or gastric and duodenal ulcer, etc;
* Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal within 14 days prior to screening;
* Concomitant therapy with any drugs with known hepatic enzyme-inducing or inhibiting agents that may change the activity of drug metabolic enzymes ，is intended to be taken in combination 28 days prior to screening or during the study period；
* Participated in another clinical research study or received any investigational products within 3 months prior to dosing;
* Presence of clinically significant abnormalities in ECG , QTcB>450ms in males,or QTcB>470ms in females;
* Any of the following diseases (including but not limited to gastrointestinal, renal, liver, neurological, hematological, endocrine, tumor, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular diseases) that are clinically significant in clinical laboratory examination or other clinical findings within 6 months prior to screening;
* Breast-feeding women or those with positive pregnancy test results;
* Subjects who should not be included in the study in the opinion of the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics | pre-dose and up to 72hours post-dose
  Tmax
Plasma pharmacokinetics | pre-dose and up to 72hours post-dose
  t1/2
Plasma pharmacokinetics | pre-dose and up to 72hours post-dose
  Cmax
Plasma pharmacokinetics | pre-dose and up to 72hours post-dose
  AUC0-∞
Plasma pharmacokinetics | pre-dose and up to 72hours post-dose
  CL/F
Number of treatment-emergent adverse events (TEAEs) and Serious Adverse Events(SAE) | up to 37days
  TEAEs will be summarized displaying the number of TEAEs along with the number and percentage of participants with at least one TEAE according to: Number of AEs, Severity and relation to study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pang Y, Li H, Chen X, Cao Y, Jiang H, Huang J, Liu Y. A phase I, single-center, randomized, open-label, three-period crossover study to evaluate the drug-drug interaction between ZSP1273 and oseltamivir in healthy Chinese subjects. Antimicrob Agents Chemother. 2025 Apr 2;69(4):e0172924. doi: 10.1128/aac.01729-24. Epub 2025 Feb 24. PMID 39992105